CLINICAL TRIAL: NCT05349669
Title: Cytokine With Jafron Haemoadsorption During Cardiopulmonary Bypass: Protocol for Randomized Controlled Report
Brief Title: Jafron Haemoadsorption During Cardiopulmonary Bypass
Acronym: JAFRONCPB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthea Hospital Bari (Other)
Responsible Party: Principal Investigator, Ignazio Condello, Principal Investigator, Anthea Hospital Bari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANTHEAHOSPITAL12022022
Record Dates: First submitted 2022-04-08; First posted 2022-04-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cytokine Release Syndrome
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CPB (No Intervention): Elective cardiopulmonary bypass (CPB) procedures with an expected time >120 minutes for each extracorporeal procedure.
- CPB with Jafron (Experimental): Elective cardiopulmonary bypass (CPB) procedures with Jafron use with an expected time >120 minutes for each extracorporealprocedure.
  Interventions: Drug: Jafron use during CPB

INTERVENTIONS:
Drug: Jafron use during CPB — Use of filter Jafron during CPB
  Arms: CPB with Jafron

SUMMARY:
Cardiopulmonary bypass (CPB) is often associated with degrees of complex inflammatory response mediated by various cytokines. This response can, in severe cases, lead to systemic hypotension and organ dysfunction. Cytokine removal might therefore improve outcomes of patients undergoing cardiac surgery. Jafron is a device designed to remove cytokine from the blood using haemoadsorption (HA). This preliminary report aims to evaluate the potential of Jafron to decrease peri-operative cytokine levels in cardiac surgery.

DETAILED DESCRIPTION:
In this context the investigators introduce the study design for multi-centre pilot randomized report in 40 patients undergoing elective CPB procedures with an expected time >120 minutes for each extracorporeal procedure. Patients will be randomly allocated to either standard of care (n = 20) or Jafron HA(n = 20) during cardiopulmonary bypass (CPB). The primary outcome will be the difference between the two groups in cytokines levels (IL-2, IL-6,TNF-α, IFN gamma) and secondary parameters (Fibrinogen, Albumin, Platelets, Hemoglobin, Hematocrit, White Blood Cells, Neutrophils,Lymphocytes, Monocytes, Eosinophils, Basophils) will measured at anaesthesia induction, at the endof CPB , Primary outcomes: hemodynamics with or without vasoconstrictors use, the mechanical ventilation (MV) (hours) time and length of stay in intensive care unit (ICU) (hours). This prospectivemulti-centre randomized controlled report will take place in two Centres: Anthea Hospital, GVMCare & Research, Bari, Italy; Virgen de la Arrixaca University Hospital, Murcia, Spain; between May 2022 and September 2022. The target population per centre will include (n=20) patients; will beallocate for each center to either standard of care (n = 10) or Jafron HA (n = 10) planned for elective cardiac surgery with increased risk of cytokine release.

ELIGIBILITY:
Inclusion Criteria :

* elective cardiac surgery under CPB
* double valve replacement or a complex surgery with an expected CPB duration > 120 min
* redo cardiac surgery

Exclusion criteria:

* end-stage renal disease (dialysis dependence)
* active infectious endocarditis
* emergency or off-pump procedure
* prescription of non-steroidal antiinflammatory medication (except for low-dose aspirin) or corticosteroids within 7 days
* enrolment in another conflicting study
* administration of human albumin during CPB

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
cytokines levels | 1 hour before start of the cardiopulmonary bypass
  IL-2, IL-6,TNF-α, IFN gamma
cytokines levels | 10 minutes after stop the cardiopulmonary bypass
  IL-2, IL-6,TNF-α, IFN gamma,
Hemodynamics supports | 10 minutes after stop of the cardiopulmonary bypass
  vasoconstrictors use or not use
Post-operative ITEMS in intensive care unit | 3 days after surgery
  mechanical ventilation (MV) (hours) time and length of stay in intensive care unit (ICU) (hours)

SECONDARY OUTCOMES:
Markers levels | 1 day before start of the cardiopulmonary bypass
  Concentration of Fibrinogen, Albumin, Platelets, Hemoglobin, Hematocrit, White Blood Cells, Neutrophils,Aptoglobin, Cell free Hemoglobin Lymphocytes, Monocytes, Eosinophils, Basophils
Markers | 1 day after stop the cardiopulmonary bypass
  Concentration of Fibrinogen, Albumin, Platelets, Hemoglobin, Hematocrit, White Blood Cells, Neutrophils,Aptoglobin, Cell free Hemoglobin Lymphocytes, Monocytes, Eosinophils, Basophils
Hemodynamics supports | 1 hour after stop the cardiopulmonary bypass
  Need of vasoconstrictors

CONTACTS AND LOCATIONS:
Locations (1):
- Anthea Hospital, Bari, Apulian, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Condello I, Morvillo JB, Fiore F, Teora V, Nasso G, Speziale G. Hemadsorption to Contain Postoperative Cell-Free Hemoglobin and Haptoglobin Preservation for Extended Cardiopulmonary Bypass Time in Cardiac Surgery for Acute Kidney Injuries Prevention. Braz J Cardiovasc Surg. 2024 May 15;39(3):e20230272. doi: 10.21470/1678-9741-2023-0272. PMID 38748856